CLINICAL TRIAL: NCT06070571
Title: Clinical Assessment of Antibacterial Anti-inflammatory Activities of Yarrow Moringa Herbal Combinations in Bucco Adhesive Films
Brief Title: Clinical Evaluation and Assesment of Ginigivitis Patients Treated by Yarrow Natural Extract in Compare to a Contro Group
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3/23
Record Dates: First submitted 2023-09-24; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Achillea millefolium flower

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Bucco-adhesive films with Yarrow and Moringa extract nanoparticles
  Interventions: Drug: Yarrow and moringa mixture
- control group (Active Comparator): Cholorohexiden oral gargles
  Interventions: Drug: Yarrow and moringa mixture

INTERVENTIONS:
Drug: Yarrow and moringa mixture — yarrow and moringa mixture nano particles loaded on buccal film

SUMMARY:
A double-blind, prospective, randomized, intra-individual comparative, single-center clinical study was conducted. Participants were placed in parallel groups, and the study was performed in the Department of Operative Dentistry and Periodontology, Dental School and Hospital, Minia university to compare the antibacterial activity of yarrow Moringa herbal combinations nanoparticles in compared to Chlorhexidine as a potential treatment for gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* a minimum of four natural uncrowned teeth in one quadrant present
* good general health
* can follow instructions

Exclusion Criteria:

* were pregnant or breastfeeding
* evidence of antibiotic use during the 4 weeks prior to the study
* were allergic to personal care/consumer products or their ingredients

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
antibacterial and anti inflammatory activities | two weeks
  scoring of erthymia and pain (no pain=0) and the other end (worst pain=10).

CONTACTS AND LOCATIONS:
Overall Officials: soad ali, PhD, Study Director — faculty of pharmacy, Deraya university
Locations (1):
- Soad A. Mohamad, Minya, Minya Governorate, Egypt